CLINICAL TRIAL: NCT07204691
Title: A SINGLE-ARM, OPEN-LABEL CLINICAL INVESTIGATION TO EVALUATE THE SAFETY AND PERFORMANCE OF DKL CROSSLINKED SODIUM HYALURONATE 20 MG/ML +LIDOCAINE 0.3% DERMAL FILLER FOR LIP AUGMENTATION
Brief Title: A Study to Evaluate the Safety and Performance of Dr Korman Laboratories' Hyaluronic Acid Filler 20 mg/mL With Lidocaine for Lip Augmentation
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Korman Laboratories Ltd. (Industry)
Collaborators: CTC Clinical Trial Consultants AB (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLSHA+L-DKL-CS001
Record Dates: First submitted 2025-09-24; First posted 2025-10-02 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Lip Augmentation
Keywords: lips; hyaluronic acid; dermal filler; esthetics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): DKL crosslinked sodium hyaluronate 20 mg/mL + Lidocaine 0.3% dermal filler (RadiaNt Soft Lidocaine)
  Interventions: Device: DKL crosslinked sodium hyaluronate 20 mg/mL + Lidocaine 0.3% dermal filler

INTERVENTIONS:
Device: DKL crosslinked sodium hyaluronate 20 mg/mL + Lidocaine 0.3% dermal filler — DKL crosslinked sodium hyaluronate 20 mg/mL + lidocaine 0.3% dermal filler is an injectable sterile, non-pyrogenic gel composed of crosslinked sodium hyaluronate of a non-animal origin and lidocaine in a phosphate-buffered saline solution.

SUMMARY:
This study will assess the safety and effectiveness of a dermal filler called DKL crosslinked hyaluronic acid 20 mg/mL with lidocaine 0.3% when injected into the lips of healthy men and women who want to have fuller lips. The change in the appearance of the lips will be checked.

DETAILED DESCRIPTION:
This is a single-arm, open-label, multi-center clinical investigation to evaluate the safety, performance, and usability of DKL crosslinked hyaluronic acid 20 mg/mL + lidocaine 0.3% for lip augmentation in healthy male and female volunteers with thin lips. Eligible participants will undergo treatment with crosslinked hyaluronic acid 20 mg/mL + lidocaine 0.3% injected into the lips for lip augmentation. Each participant will act as his/her own control. The improvement in lip appearance over time will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Review and sign the IEC-approved Informed Consent Form (ICF) prior to any clinical investigation-related procedures being performed. In addition, the subject will be asked to provide a separate release for the use of their photographs in publications and the clinical investigation report (CIR). The subject has a right to refuse the photo release without jeopardizing their eligibility to participate in the clinical investigation.
2. Healthy male or female subject aged 18 inclusive, at the time of screening.
3. Has both an upper and lower lip that are very thin, or thin on the LFGS, and desires at least a 1-point improvement in LFGS score in either lip.
4. Female of childbearing potential (sexually active and not sterile nor postmenopausal for at least 1 year) should have a urine pregnancy test evaluated as negative on the day of enrollment and agree to use a reliable method of contraception for the duration of the clinical investigation (effective birth control measures include sexual abstinence, combined [estrogen and progestogen containing] hormonal contraception associated with inhibition of ovulation [oral, intravaginal, transdermal], progestogen-only hormonal contraception associated with inhibition of ovulation [oral, injectable, implantable], intrauterine device [IUD] or intrauterine hormone-releasing system [IUS] and/or condom with spermicide).
5. The subject has an adequate understanding of the local language to understand verbal and written subject information and is willing to comply with the clinical investigation requirements.

Exclusion Criteria:

1. History of any clinically significant disease or disorder which, in the opinion of the Investigator, may either put the subject at risk because of participation in the clinical investigation or influence the results or the subject's ability to participate in the clinical investigation.
2. Any clinically significant illness, medical/surgical procedure, or trauma within 4 weeks prior to the first administration of the investigational device.
3. Subjects with epilepsy.
4. History of streptococcal disease (such as recurrent sore throats), rheumatic fever or acute rheumatic fever.
5. Current smokers or users of nicotine products. Irregular use of nicotine (e.g., smoking, snus/nicotine pouches, snuffing, chewing tobacco) less than 3 times/week before the screening visit is allowed.
6. Known hypersensitivity to HA and/or to gram-positive bacterial proteins, as HA.
7. History of allergy, anaphylaxis, or hypersensitivity to injectable HA products, local anesthetics of the amide-type such as lidocaine, or latex, or is planning to undergo desensitization therapy during the clinical investigation.
8. Has lip tattoos, piercings, facial hair, tissue damage/malformation in the mouth (e.g., due to snus/nicotine pouch use) or scars that would interfere with visualization of the lips and perioral area for the effectiveness assessments.
9. Has abnormal lip function, with an inability to effectively sip water through a straw.
10. Has abnormal lip sensation, with an inability to feel a 0.4G monofilament or a cotton wisp at any site on the lip.
11. Has moderate or severe abnormal lip asymmetry.
12. Has any mass-formation on the lip.
13. Has dentures or any device covering all or part of the upper palate, and/or severe malocclusion or dentofacial or maxillofacial deformities as judged by the Treating Investigator. Subjects planning to undergo extensive dental procedures such as dental implants, multiple tooth extractions, or oral surgery should not participate. Minor dental procedures such as teeth cleaning and repair of caries are not exclusionary.
14. Has used ANY lip filling agents within 12 months of clinical investigation enrollment (HA products, collagen-based products, etc.).
15. Has used permanent and/or semi-permanent lip filling agents (e.g., silicone, collagen, calcium).
16. Has used any lip-plumping products or devices within 10 days before enrollment or is planning to use such products during the clinical investigation.
17. Has begun using any over-the-counter (OTC) or prescription oral or topical anti-wrinkle products for the lips or around the mouth within 90 days before enrollment or is planning to begin using such products during the clinical investigation (subjects who have been on a stable regimen of such products for at least 90 days are eligible for the clinical investigation and must continue their regimen throughout the clinical investigation.)
18. Is on an ongoing regimen of anti-coagulation therapy (e.g., warfarin), thrombolytics, or inhibitors of platelet aggregation or non-steroidal anti-inflammatory drugs (NSAIDs, e.g., aspirin, ibuprofen) or other substances known to increase coagulation time (e.g., herbal supplements with garlic or ginkgo) within 10 days of undergoing clinical investigation device injections.
19. Has a history or presence of bleeding disorders.
20. Has used systemic corticosteroids or immunosuppressive medications within 30 days prior to treatment.
21. Is on a concurrent regimen of lidocaine or structurally related local anesthetics (e.g., bupivacaine).
22. Has an active inflammation (skin eruptions such as cysts, pimples, rashes, or hives), infection, cancerous or pre-cancerous lesion, or unhealed wound on the face.
23. Has a history of known susceptibility to keloid formation or hypertrophic scars.
24. Has active herpes labialis lesions at the time of injections. Subjects with a history of herpes labialis who have had four or more outbreaks in the 12 months prior to enrollment are also excluded even in the absence of lesions at the baseline visit.
25. Subjects who are pregnant, lactating, or planning to become pregnant at any time during the clinical investigation.
26. History of alcohol or drug abuse or excessive intake of alcohol, as judged by the Investigator.
27. Has received any investigational device within 30 days prior to clinical investigation enrollment or is planning to participate in another investigation during the course of this clinical investigation.
28. Is an employee (or a relative of an employee) of the Monitor or contract research organization (CRO) responsible for conducting the clinical investigation, the Sponsor, or a Sponsor representative.
29. The Investigator considers the subject unlikely to comply with clinical investigation procedures, restrictions, and requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2025-09-24 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Change in Lip Fullness Grading Scale (LFGS) score from baseline to 8 weeks after treatment. | Baseline (prior to treatment) to Week 8
  The LFGS is a validated 5-point photonumeric rating scale that quantifies lip fullness on a scale ranging from very thin (0) to full (4).

SECONDARY OUTCOMES:
Change in Lip Fullness Grading Scale (LFGS) score from baseline to 4, 12, 16, 24 and 48 weeks. | Baseline (prior to treatment) to Week 4, 12, 16, 24 and 48.
  The LFGS is a validated 5-point photonumeric rating scale that quantifies lip fullness on a scale ranging from very thin (0) to full (4).
The percentage of subjects who had an improvement of at least one point in the LFGS score from baseline to 4, 8, 12, 16, 24, and 48 weeks. | Baseline (prior to treatment) to Week 4, 8, 12, 16, 24, and 48.
  The LFGS is a validated 5-point photonumeric rating scale that quantifies lip fullness on a scale ranging from very thin (0) to full (4).
Investigator-rated aesthetic improvement in appearance according to the Global Aesthetic Improvement Scale (GAIS) at 4, 8, 12, 16, 24, and 48 weeks after the initial treatment. | Baseline (prior to treatment) to Week 4, 8, 12, 16, 24, and 48.
  The GAIS is a 5-point scale rating global aesthetic improvement in appearance. The rating categories range from 'worse' to 'very much improved'.
Percentage of responders defined as at least "improved" (improved, much improved, very much improved) as assessed by the Investigator-rated GAIS at 4, 8, 12, 16, 24, and 48 weeks after the initial treatment. | Baseline (prior to treatment) to Week 4, 8, 12, 16, 24, and 48.
  The GAIS is a 5-point scale rating global aesthetic improvement in appearance. The rating categories range from 'worse' to 'very much improved'.
Subject-rated aesthetic improvement in appearance according to GAIS at 4, 8, 12, 16, 24, and 48 weeks after the initial treatment. | Baseline (prior to treatment) to Week 4, 8, 12, 16, 24, and 48.
  The GAIS is a 5-point scale rating global aesthetic improvement in appearance. The rating categories range from 'worse' to 'very much improved'.
Percentage of responders defined as at least "improved" (improved, much improved, very much improved) as assessed by subject-rated GAIS at 4, 8, 12, 16, 24, and 48 weeks after the initial treatment. | Baseline (prior to treatment) to Week 4, 8, 12, 16, 24, and 48.
  The GAIS is a 5-point scale rating global aesthetic improvement in appearance. The rating categories range from 'worse' to 'very much improved'.
The intensity of pain during the initial injection and touch-up, evaluated on a numerical rating scale (NRS) ranging from 1 (no pain at all) to 10 (worst pain ever possible). | Baseline (initial treatment), 4 weeks (touch-up, if applicable)
  The NRS measures the intensity of pain from 1 (no pain at all) to 10 (worst pain ever possible).
Frequency, intensity, and duration of pre-defined expected post-treatment events collected using a subject diary for 14 days post-treatment. | From baseline to Week 2; if touch up is done: From Week 4 to Week 6
  The frequency, intensity, and duration of pre-defined expected post-treatment events collected using a subject diary.
Frequency, intensity, and duration of adverse events (AEs) throughout the clinical investigation and up to 48 weeks. | Baseline to Week 48
  The frequency, intensity, and duration of adverse events.
Incidence of device deficiencies (DDs). | Baseline to Week 4
  The incidence of DDs.
Lip function, sensation, texture, firmness, and movement/function, before injection and at 4, 8, 12-, 16-, 24-, and 48 weeks post-baseline. | Baseline to Week 4, 8, 12, 16, 24, and 48.
  Lip function, sensation, texture, firmness, and movement/function will be assessed as normal or abnormal.
Subject satisfaction using the validated FACE-Q scales: • Satisfaction with Lips • Satisfaction with Outcome | Baseline to Week 4, 8, 12, 16, 24, and 48 (Satisfaction with outcome will not be assessed at baseline).
  Satisfaction with Lips is a 10-item scale measures the appearance of the lips with items that ask about size, shape, and fullness, as well as how their lips suit their face and how the lips look when smiling. The answers range from very dissatisfied (1), to very satisfied (4).
  Satisfaction with Outcome is a 6-item scale measures satisfaction with the result of a facial procedure. The answers range from agree (1) to disagree (4).
Investigator-reported usability of the device | Week 4 (after completing the treatment of all subjects)
  A usability questionnaire will be completed by each of the Treating Investigators.

CONTACTS AND LOCATIONS:
Locations (2):
- Sweden (2):
  - Clinical Trial Consultants AB (CTC) GoCo, Mölndal
  - CTC Stockholm, Solna

IPD SHARING:
Plan to Share IPD: No